CLINICAL TRIAL: NCT03657758
Title: Lesional Evaluation of High Risk Patients With Neoatherosclerosis Treated With Rosuvastatin and Eicosapentaenoic Acid Using OCT
Brief Title: Lesional Evaluation of High Risk Patients With Neoatherosclerosis Treated With Rosuvastatin and Eicosapentaenoic Acid Using Optical Coherence Tomography(OCT)[LINK IT TWO]
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, Senior Lecturer, Kobe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300027
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: eicosapentaenoic acid; OCT; neoatherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPA and statin therapy group (Active Comparator): After randomization, patients with combination therapy start EPA (1800mg/day) and high dose rosuvastatin (10mg/day) for ９ months.
  Interventions: Drug: EPA and rosuvastatin
- High dose statin therapy group (Active Comparator): After randomization, patients with high dose statin therapy start high dose rosuvastatin (10mg/day) for ９ months.
  Interventions: Drug: High dose rosuvastatin
- low dose statin therapy group (No Intervention): After randomization, patients with low dose statin therapy take low dose rosuvastatin (5mg/day) for ９ months.

INTERVENTIONS:
Drug: EPA and rosuvastatin — To take EPA (1800mg/day) and high dose rosuvastatin (10mg/day) for ９ months.
  Arms: EPA and statin therapy group
Drug: High dose rosuvastatin — To take high dose rosuvastatin (10mg/day) for ９ months.
  Arms: High dose statin therapy group

SUMMARY:
This study aim is to evaluate the additional effect of eicosapentaenoic acid and dose up effect of rosuvastatin for neoatherosclerosis in coronary artery disease patients.

DETAILED DESCRIPTION:
Eicosapentaenoic acid and statin therapy prevents cardiovascular events. However, the impact of these treatment in patients with in-stent neoatherosclerosis has not been clarified.

So, the investigators conducted LINK IT study. This study showed that eicosapentaenoic acid(EPA) and rosuvastatin therapy improve lipid index in patients compared with rosuvastatin alone therapy.

However, it was insufficient to directly evaluate the efficacy of additional effect of EPA for neoatherosclerosis. Because, statin dose of two groups was different and type of stent was variety.

Therefore, the investigators designed a new prospective, randomized OCT study. The OCT operators randomly assigned 75 patients who were detected neoatherosclerosis on follow-up OCT examination after implanted everolimus eluting stent to three groups; 5mg/day of rosuvastatin therapy (low dose statin therapy group) or 10mg/day of rosuvastatin therapy (high dose statin therapy group) or 10mg/day of rosuvastatin and 1800mg/day of eicosapentaenoic acid therapy (EPA and statin therapy group). Serial coronary angiography and OCT were performed at 9 months after baseline OCT procedure.

This study aim is to evaluate the additional effect of eicosapentaenoic acid and dose up effect of rosuvastatin for neoatherosclerosis in coronary artery disease patients by comparing 3 groups.

ELIGIBILITY:
Inclusion Criteria:

1. over 20 years
2. Patients implanted everolimus-eluting stent(EES) neoatherosccrelosis with neoatherosclerosis by OCT
3. LDL is or less than 100 mg/dl after ingesting 5 mg/day of rosuvastatin

Exclusion Criteria:

1. Patients taking omega 3 fatty acid before randomization
2. Patients allergic to rosuvastatin or eicosapentaenoic acid
3. Patients with a history of hemorrhagic stroke
4. Patients taking anti cancer agent
5. Patients undergoing LDL apheresis
6. Patients with severe liver disease or severe kidney disease
7. Patients who conflict with any of the warnings or contraindications listed in the domestic package insert of rosuvastatin
8. Patients who conflict with any of the warnings or contraindications listed in the domestic package insert of eicosapentaenoic acid
9. Patients performed percutaneous coronary intervention with restenosis of target lesion
10. Pregnant women or patients with possibility of Pregnancy or nursing woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-09-17 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
The change in lipid index | 9 months
  mean lipid arc ✕ lipid length

SECONDARY OUTCOMES:
MACE | 9 months
  Major cerebro-cardiovascular events（Nonfatal stroke, Nonfatal myocardial infarction, cardiovascular death)
The change in minimum lumen area | 9 months
  OCT parameter
The change in average neointimal thickness | 9 months
  OCT parameter
The change in lipid arc | 9 months
  OCT parameter
The change in lipid length | 9 months
  OCT parameter
The change in thin cap fibroatheroma | 9 months
  OCT parameter
The change in macrophage grade | 9 months
  OCT parameter
The change in plaque volume | 9 months
  Near infrared spectroscopy intravascular ultrasound(NIRS-IVUS) parameter
The change in max Lipid-core burden index | 9 months
  NIRS-IVUS parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Kobe University Graduate School of Medicine, Department of Cardiology, Kobe, Hyōgo, Japan